CLINICAL TRIAL: NCT07093814
Title: A Phase I/II Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of VRT106 for Injection in Patients With Recurrent/Progressive Glioblastoma
Brief Title: A Study of VRT106 for Injection in Patients With Recurrent/Progressive Glioblastoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangzhou Virotech Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRT106-CN02（INVIGOR-101）
Record Dates: First submitted 2025-07-15; First posted 2025-07-30 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma
Keywords: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VRT106 (Experimental): VRT106 will be administered intravenously
  Interventions: Drug: VRT106

INTERVENTIONS:
Drug: VRT106 — VRT106,intravenous

SUMMARY:
This study is an open-label, single-arm Phase I/II clinical trial with the primary objective of evaluating the safety, tolerability, and efficacy of VRT106 in patients with recurrent/progressive glioblastoma.

DETAILED DESCRIPTION:
This study is an open-label, single-arm Phase I/II clinical trial comprising two parts: Phase I and Phase II. Phase I is a dose-escalation phase, with the primary objective of assessing the safety and tolerability of VRT106 at escalating doses in subjects with recurrent/progressive glioblastoma and confirming the Recommended Phase II Dose (RP2D). Phase II is a dose-expansion phase, in which subjects will receive VRT106 at the RP2D dose level, aiming to further evaluate the efficacy and safety of VRT106 in subjects with recurrent/progressive glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in the clinical study; fully understand and be informed about the study and sign the ICF; and are willing to follow and have the ability to complete all trial procedures.
* Males and females are aged at 18-70 years (including borderline values) at the time of signing the ICF, male or female.
* Diagnosed with recurrent/progressive glioblastoma.
* Karnofsky Performance Status (KPS) score ≥60 within 28 days prior to the first administration of the study drug.
* An expected survival time of≥3 months.
* Have sufficient organ function.
* Female patients of childbearing potential must have a negative serum pregnancy test result within 7 days prior to the first use of the study drug (if a false-positive pregnancy test result is due to non-pregnancy factors such as illness, further testing via ultrasound or other methods is required, and the investigator must confirm the absence of pregnancy before enrollment).
* Subjects of childbearing potential (males and females) agree to use effective birth control with their partner from signing informed consent to at least 90 days after the last dose.

Exclusion Criteria:

* Patients with extracranial metastases.
* Previously received treatment with oncolytic viruses, gene therapy.
* Subject has received treatment with other unlisted clinical investigational drugs/devices within 4 weeks prior to the first dose of VRT106.
* Subject is known to have an allergic reaction to any of the components of VRT106.
* Patients who can't have a cranial MRI scan.
* Women who are breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of escalating doses of VRT106 in Patients with recurrent/progressive glioblastoma | About 2 years
  To evaluate the safety and tolerability of VRT106 in patients with recurrent/progressive glioblastoma and to explore the maximum tolerated dose (MTD)/multiple ascending dose (MAD)/optimal biologically active dose (OBD) and/or the recommended phase 2 dose(RP2D), which will provide a recommended dose for subsequent clinical trials. The specific outcome indicator data that need to be evaluated and collected include: adverse event, physical examinations, vital signs, clinical laboratory tests (including blood routine, blood biochemistry.urine routine, coagulation function), Eastern Cooperative Oncology Group (ECOG) performance status, twelve-lead electrocardiogram(ECG) and concomitant medication assessments.

SECONDARY OUTCOMES:
Overall survival | About 2 years
  Time from initial administration to death
Objective response rate | About 2 years
  Objective response rate assessed according to the Neuro-Oncology Response Evaluation Criteria, complete response (CR) + partial response (PR)
Distribution and shedding of VRT106 virus | About 2 years
  Concentration of VRT106 virus in blood
Overall survival rate | About 2 years
  Overall survival rates at 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chengcheng Guo, Principal Investigator — Sun Yat-sen University
Locations (11):
- China (11):
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - Sanbo Brain Hospital Capital Medical University, Beijing, Beijing Municipality
  - The Cancer Hospital Affiliated to Chongqing University, Chongqing, Chongqing Municipality
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Tangdu Hospital of Air Force Medical University of the PLA, Xi’an, Shanxi
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang